CLINICAL TRIAL: NCT01006772
Title: Rehabilitation of Early Stroke Patients Using a Custom-made Solid Ankle-foot Orthosis: a Randomised Controlled Trial
Brief Title: Rehabilitation of Early Stroke Patients Using an AFO: an RCT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Strathclyde (Other)
Responsible Party: Enrica Papi (Bioengineering Department, University of Strathclyde), University of Strathclyde
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHILIPROWE1
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2009-11

CONDITIONS: Stroke; Hemiplegia
Keywords: Stroke; Ankle Foot Orthosis; Walking Speed; Gait; Rehabilitation; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Control group patients receive usual clinical practice provided by Stroke Unit at Stobhill Hospital in Glasgow. They receive physiotherapy and early mobilisation as deemed appropriate to treat their oown impairments.
- Experimental group (Experimental): Intervention Group patients receive custom made solid ankle foot orthosis (AFO)treatment.
  Interventions: Other: Solid Ankle Foot Orthosis

INTERVENTIONS:
Other: Solid Ankle Foot Orthosis — Polypropylene (homopolymer) AFO with carbon fiber reinforcements is provided to experimental group patients as an adjunct therapy to conventional physical therapy.
  Other Names: Solid Ankle foot orthosis users
  Arms: Experimental group

SUMMARY:
Stroke is a major cause of disabilities worldwide. Stroke survivors commonly exhibit walking defects which lead to an altered, slow speed and asymmetric gait pattern. The main aims of rehabilitation are to enhance recovery of movement control and regain walking ability. Ankle-foot orthoses (AFOs), braces which encompass the foot and ankle joint extending to a point below the knee, are commonly prescribed to address ambulation impairments in stroke patients. Their main function is to support the foot and allow a subject to walk safely with a gait approaching normality. This project will aim to evaluate the early provision of AFOs as an adjunct to standard physiotherapy on the walking ability of stroke survivors. Usual rehabilitation practice will be the control condition. Participants will be recruited from the stroke unit of Stobhill Hospital in Glasgow. They will be randomised into two groups. Participants allocated in the control group will receive usual clinical practice as per routine for stroke patients. The intervention group will receive custom made solid AFOs as an adjunct. They will be provided with three AFOs, one for use during rehabilitation and two which will be used only during the outcome assessment sessions for research purposes. The intervention phase will last 24 weeks. Gait analysis will be performed three times for each participant (at baseline, 12 and 24 weeks after enrolment) in the biomechanical laboratory of Strathclyde University. During these sessions force and movement data of patients walking will be recorded. Fortnightly time and distance factors of gait will be measured and a battery of functional tasks will be performed in the physiotherapy gym of the hospital using a simple video camera and a grid lino-mat. During all assessments participants with an AFO will be asked to walk with and without the AFO provided.

ELIGIBILITY:
Inclusion Criteria:

* 7 days to 8 weeks after ischemic or haemorrhagic stroke, medically stable, age range between 18 and 90 years, gastrocnemius shortening with plantarflexion contracture (5 degrees of plantarflexion or greater), capable of full correction of subtalar joint, no loss of skin integrity over the lower limb, no severe cognitive impairments, sufficient communication to follow the instructions in the trial data collection procedures (follow a single one step command).

Exclusion Criteria:

* Inability to follow simple instructions or to give informed consent, unstable angina, cardiac risks, pain related to walking, severe spasticity, the need for two assistants while walking, severe proprioceptive sensory impairment, soleus contracture which prevents casting for the AFO at 90 degrees , flexion contracture of hip musculature (greater than 10 degrees hip flexion).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-04 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
walking speed | every 2 weeks

SECONDARY OUTCOMES:
Ground reaction force value and alignment | every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Rowe, PhD, BSc, MISB, Study Director — University of Strathclyde
Locations (1):
- Bioengineering Departent (University of Strathclyde), Glasgow, United Kingdom